CLINICAL TRIAL: NCT01888497
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, CROSS-OVER, PLACEBO-CONTROLLED, SINGLE DOSE, CLINICAL TRIAL TO ASSESS THE NEXT-DAY RESIDUAL EFFECTS OF GABAPENTIN, DIPHENHYDRAMINE AND TRIAZOLAM ON SIMULATED DRIVING PERFORMANCE IN NORMAL VOLUNTEERS
Brief Title: Next-Day Residual Effects of Gabapentin, Diphenhydramine and Triazolam on Simulated Driving Performance in Normal Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A9451178
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Sleeplessness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Gabapentin; Diphenhydramine; Triazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Experimental)
  Interventions: Drug: Gabapentin
- Arm B (Experimental)
  Interventions: Drug: Diphenhydramine citrate
- Arm C (Active Comparator)
  Interventions: Drug: Triazolam
- Arm D (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — 250 mg, oral, prior to bedtime on the night before performance testing
  Arms: Arm A
Drug: Diphenhydramine citrate — 76 mg, oral, prior to bedtime on the night before performance testing
  Arms: Arm B
Drug: Triazolam — 0.5 mg, oral, prior to bedtime on the night before performance testing
  Arms: Arm C
Drug: Placebo — Oral, prior to bedtime on the night before performance testing
  Arms: Arm D

SUMMARY:
This study will examine the next-day residual effects of a nighttime dose of gabapentin 250 mg, diphenhydramine citrate 76 mg and triazolam 0.5 mg compared to placebo and each other on simulated driving performance in normal volunteer subjects. It will also examine other measures of next-day performance and next-day sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females of non-childbearing potential, 25-55 years of age
* Valid driver's license

Exclusion Criteria:

* Psychiatric disorder
* Recent history of clinically significant neurological disorder, such as seizures, stroke, multiple sclerosis, or head trauma
* Recent histroy or current treatment for sleep disorder

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2013-12-14 (Actual); Study Completion 2013-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Baptist Sleep Centers, LLP, South Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - NeuroTrials Research Sleep Lab, Atlanta, Georgia
  - NeuroTrials Research, Inc., Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451178&StudyName=Next-Day%20Residual%20Effects%20of%20Gabapentin%2C%20Diphenhydramine%20and%20Triazolam%20on%20Simulated%20Driving%20Performance%20in%20Normal%20Volunteers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, all participants were screened for simulator sickness and underwent standardized training on the driving simulator to ensure that participants fully understood how to perform the tests, were comfortable, and attained a stable level of performance on the various performance-based measures.
Groups:
- Diphenhydramine Citrate, Gabapentin, Placebo, Triazolam: A single dose of 1 diphenhydramine citrate 76 milligram (mg) capsule and 2 placebo tablets orally in first intervention period followed by a single dose of 1 gabapentin 250 mg capsule and 2 placebo tablets orally in second intervention period, then a single dose of 1 placebo capsule and 2 placebo tablets orally in third intervention period and then a single dose of 2 triazolam 0.25 mg tablets (equivalent to triazolam 0.5 mg) and 1 placebo capsule orally in fourth intervention period. Each intervention period consisted of dosing day on which the study treatment was administered at night followed by testing day. A washout period of 7 to 14 days was maintained between each intervention period.
- Gabapentin, Triazolam, Diphenhydramine Citrate, Placebo: A single dose of 1 gabapentin 250 mg capsule and 2 placebo tablets orally in first intervention period followed by a single dose of 2 triazolam 0.25 mg tablets (equivalent to triazolam 0.5 mg) and 1 placebo capsule orally in second intervention period then a single dose of 1 diphenhydramine citrate 76 mg capsule and 2 placebo tablets orally in third intervention period and then a single dose of 1 placebo capsule and 2 placebo tablets orally in fourth intervention period. Each intervention period consisted of dosing day on which the study treatment was administered at night followed by testing day. A washout period of 7 to 14 days was maintained between each intervention period.
- Triazolam, Placebo, Gabapentin, Diphenhydramine Citrate: A single dose of 2 triazolam 0.25 mg tablets (equivalent to triazolam 0.5 mg) and 1 placebo capsule orally in first intervention period followed by 1 placebo capsule and 2 placebo tablets orally in second intervention period then a single dose of 1 gabapentin 250 mg capsule and 2 placebo tablets orally in third intervention period and then a single dose of 1 diphenhydramine citrate 76 mg capsule and 2 placebo tablets orally in fourth intervention period. Each intervention period consisted of dosing day on which the study treatment was administered at night followed by testing day. A washout period of 7 to 14 days was maintained between each intervention period.
- Placebo, Diphenhydramine Citrate, Triazolam, Gabapentin: A single dose of 1 placebo capsule and 2 placebo tablets orally in first intervention period followed by a single dose of 1 diphenhydramine citrate 76 mg capsule and 2 placebo tablets orally in second intervention period then a single dose of 2 triazolam 0.25 mg tablets (equivalent to triazolam 0.5 mg) and 1 placebo capsule orally in third intervention period and then a single dose of gabapentin 250 mg capsule and 2 placebo tablets orally in fourth intervention period. Each intervention period consisted of dosing day on which the study treatment was administered at night followed by testing day. A washout period of 7 to 14 days was maintained between each intervention period.
Period: First Intervention Period
Arm/Group | Diphenhydramine Citrate, Gabapentin, Placebo, Triazolam | Gabapentin, Triazolam, Diphenhydramine Citrate, Placebo | Triazolam, Placebo, Gabapentin, Diphenhydramine Citrate | Placebo, Diphenhydramine Citrate, Triazolam, Gabapentin
Started | 13 | 14 | 15 | 17
Completed | 13 | 14 | 15 | 17
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Diphenhydramine Citrate, Gabapentin, Placebo, Triazolam | Gabapentin, Triazolam, Diphenhydramine Citrate, Placebo | Triazolam, Placebo, Gabapentin, Diphenhydramine Citrate | Placebo, Diphenhydramine Citrate, Triazolam, Gabapentin
Started | 13 | 14 | 15 | 17
Completed | 13 | 14 | 14 | 16
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Period: Second Intervention Period
Arm/Group | Diphenhydramine Citrate, Gabapentin, Placebo, Triazolam | Gabapentin, Triazolam, Diphenhydramine Citrate, Placebo | Triazolam, Placebo, Gabapentin, Diphenhydramine Citrate | Placebo, Diphenhydramine Citrate, Triazolam, Gabapentin
Started | 13 | 14 | 14 | 16
Completed | 13 | 14 | 14 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Diphenhydramine Citrate, Gabapentin, Placebo, Triazolam | Gabapentin, Triazolam, Diphenhydramine Citrate, Placebo | Triazolam, Placebo, Gabapentin, Diphenhydramine Citrate | Placebo, Diphenhydramine Citrate, Triazolam, Gabapentin
Started | 13 | 14 | 14 | 16
Completed | 13 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Third Intervention Period
Arm/Group | Diphenhydramine Citrate, Gabapentin, Placebo, Triazolam | Gabapentin, Triazolam, Diphenhydramine Citrate, Placebo | Triazolam, Placebo, Gabapentin, Diphenhydramine Citrate | Placebo, Diphenhydramine Citrate, Triazolam, Gabapentin
Started | 13 | 14 | 14 | 14
Completed | 13 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | Diphenhydramine Citrate, Gabapentin, Placebo, Triazolam | Gabapentin, Triazolam, Diphenhydramine Citrate, Placebo | Triazolam, Placebo, Gabapentin, Diphenhydramine Citrate | Placebo, Diphenhydramine Citrate, Triazolam, Gabapentin
Started | 13 | 14 | 14 | 14
Completed | 13 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention Period
Arm/Group | Diphenhydramine Citrate, Gabapentin, Placebo, Triazolam | Gabapentin, Triazolam, Diphenhydramine Citrate, Placebo | Triazolam, Placebo, Gabapentin, Diphenhydramine Citrate | Placebo, Diphenhydramine Citrate, Triazolam, Gabapentin
Started | 13 | 14 | 14 | 14
Completed | 13 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all randomized participants who received at least 1 dose of investigational product and provided any data post-randomization.
Groups:
- Entire Study Population: All participants randomized to receive diphenhydramine citrate first, gabapentin first, triazolam first or placebo first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Standard Deviation of Lateral Position (SDLP)
Description: Driving performance assessment for the participants were measured by simulated driving test using Cognitive Research Corporation Driving Simulator (CRCDS-MiniSim). The assessment was performed after 45 minutes of awakening from approximately 6.5 hours of sleep on testing day (after 7.25 hours of study drug administration). SDLP was used to assess driver's ability to track their lane and was the standard deviation of lane positions through the entire drive.
Time Frame: 7.25 hours post-dose
Population: ITT population included all randomized participants who received at least 1 dose of investigational product and provided any data post-randomization.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Groups:
- Placebo: A single dose of 1 placebo capsule and 2 placebo tablets orally in one of the four intervention periods.
- Gabapentin: A single dose of 1 gabapentin 250 mg capsule and 2 placebo tablets orally in one of the four intervention periods.
- Diphenhydramine Citrate: A single dose of 1 diphenhydramine citrate 76 mg capsule and 2 placebo tablets orally in one of the four intervention periods.
- Triazolam: A single dose of 2 triazolam 0.25 mg tablets (equivalent to triazolam 0.5 mg) and 1 placebo capsule orally in one of the four intervention periods.
Arm/Group | Placebo | Gabapentin | Diphenhydramine Citrate | Triazolam
Number analyzed (Participants) | 58 | 55 | 57 | 56
centimeter (cm) | 33.2 (8.0) | 34.2 (10.0) | 35.4 (8.9) | 47.4 (12.0)
Statistical Analysis 1: Comparison: Placebo vs Triazolam; For primary endpoint sequential order of testing: triazolam versus (vs) placebo; gabapentin vs placebo; diphenhydramine citrate vs gabapentin; diphenhydramine citrate vs placebo. If comparison at preceding step was significant, only then subsequent comparisons were considered significant; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum test — Statistical comparison was performed at a two-sided significance level of 0.05; Hodges-Lehman estimate = 13.82, 95% CI 2-sided [10.85 to 17.40] — Hodges-Lehman estimate of treatment difference was reported
Statistical Analysis 2: Comparison: Placebo vs Gabapentin; For primary endpoint sequential order of testing: triazolam vs placebo; gabapentin vs placebo; diphenhydramine citrate vs gabapentin; diphenhydramine citrate vs placebo. If comparison at preceding step was significant, only then subsequent comparisons were considered significant; Test type: Non-Inferiority or Equivalence — For gabapentin versus placebo comparison, the non-inferiority margin for upper limit of 95 percent (%) confidence interval (CI) was 2.4 cm; Hodges-Lehman estimate = 0.55, 95% CI 2-sided [-0.66 to 2.33] — Hodges-Lehman estimate of treatment difference was reported
Statistical Analysis 3: Comparison: Gabapentin vs Diphenhydramine Citrate; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.134, Wilcoxon Rank Sum test — Statistical comparison was performed at a two-sided significance level of 0.05; Hodges-Lehman estimate = 1.02, 95% CI 2-sided [-0.39 to 2.51] — Hodges-Lehman estimate of treatment difference was reported
Statistical Analysis 4: Comparison: Placebo vs Diphenhydramine Citrate; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum test — Statistical comparison was performed at a two-sided significance level of 0.05; Hodges-Lehman estimate = 2.37, 95% CI 2-sided [1.01 to 3.98] — Hodges-Lehman estimate of treatment difference was reported

2. Secondary Outcome: Speed Deviation
Description: Driving performance assessment for the participants were measured by simulated driving test using Cognitive Research Corporation Driving Simulator (CRCDS-MiniSim). The assessment was performed after 45 minutes of awakening from approximately 6.5 hours of sleep on testing day (after 7.25 hours of study drug administration). Standard deviation of speed was reported in the outcome measure.
Time Frame: 7.25 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters per second (m/sec)
Arm/Group | Placebo | Gabapentin | Diphenhydramine Citrate | Triazolam
Number analyzed (Participants) | 58 | 55 | 57 | 56
meters per second (m/sec) | 0.9 (0.3) | 0.9 (0.3) | 1.0 (0.3) | 1.3 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Triazolam; For secondary endpoint sequential order of testing: triazolam vs placebo; gabapentin vs placebo; diphenhydramine citrate vs gabapentin; diphenhydramine citrate vs placebo. If comparison at preceding step was significant, only then subsequent comparisons were considered significant; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum test — Statistical comparison was performed at a two-sided significance level of 0.05; Hodges-Lehman estimate = 0.36, 95% CI 2-sided [0.26 to 0.47] — Hodges-Lehman estimate of treatment difference was reported
Statistical Analysis 2: Comparison: Placebo vs Gabapentin; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — For gabapentin versus placebo comparison, the non-inferiority margin for upper limit of 95% CI was 0.1 m/sec; Hodges-Lehman estimate = -0.01, 95% CI 2-sided [-0.07 to 0.05] — Hodges-Lehman estimate of treatment difference was reported
Statistical Analysis 3: Comparison: Gabapentin vs Diphenhydramine Citrate; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.012, Wilcoxon Rank Sum test — Statistical comparison was performed at a two-sided significance level of 0.05; Hodges-Lehman estimate = 0.07, 95% CI 2-sided [0.02 to 0.12] — Hodges-Lehman estimate of treatment difference was reported
Statistical Analysis 4: Comparison: Placebo vs Diphenhydramine Citrate; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.014, Wilcoxon Rank Sum test — Statistical comparison was performed at a two-sided significance level of 0.05; Hodges-Lehman estimate = 0.06, 95% CI 2-sided [0.01 to 0.12] — Hodges-Lehman estimate of treatment difference was reported

3. Secondary Outcome: Lane Exceedance
Description: Driving performance assessment for the participants were measured by simulated driving test using Cognitive Research Corporation Driving Simulator (CRCDS-MiniSim). The assessment was performed after 45 minutes of awakening from approximately 6.5 hours of sleep on testing day (after 7.25 hours of study drug administration). Mean lanes excursed/exceeded was reported in the outcome measure.
Time Frame: 7.25 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lanes exceeded
Arm/Group | Placebo | Gabapentin | Diphenhydramine Citrate | Triazolam
Number analyzed (Participants) | 58 | 55 | 57 | 56
lanes exceeded | 37.8 (45.9) | 46.7 (58.5) | 52.4 (62.0) | 147.7 (113.6)
Statistical Analysis 1: Comparison: Placebo vs Triazolam; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum test — Statistical comparison was performed at a two-sided significance level of 0.05; Hodges-Lehman estimate = 103.25, 95% CI 2-sided [72.00 to 130.50] — Hodges-Lehman estimate of treatment difference was reported
Statistical Analysis 2: Comparison: Placebo vs Gabapentin; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — For gabapentin versus placebo comparison, the non-inferiority margin for upper limit of 95% CI was 8 lanes; Hodges-Lehman estimate = 5.00, 95% CI 2-sided [-4.00 to 16.50] — Hodges-Lehman estimate of treatment difference was reported
Statistical Analysis 3: Comparison: Gabapentin vs Diphenhydramine Citrate; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.213, Wilcoxon Rank Sum test — Statistical comparison was performed at a two-sided significance level of 0.05; Hodges-Lehman estimate = 3.00, 95% CI 2-sided [-3.00 to 9.00] — Hodges-Lehman estimate of treatment difference was reported
Statistical Analysis 4: Comparison: Placebo vs Diphenhydramine Citrate; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.003, Wilcoxon Rank Sum test — Statistical comparison was performed at a two-sided significance level of 0.05; Hodges-Lehman estimate = 11.00, 95% CI 2-sided [4.00 to 20.50] — Hodges-Lehman estimate of treatment difference was reported

ADVERSE EVENTS:
Description: Same event may appear as adverse event (AE) and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as nonserious in another participant or 1 participant may have experienced both serious and nonserious event during study. Safety population was evaluated.
Arm/Group | Placebo | Gabapentin | Diphenhydramine Citrate | Triazolam
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/55 | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 3/58 | 2/55 | 3/57 | 10/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=58) | Gabapentin (N=55) | Diphenhydramine Citrate (N=57) | Triazolam (N=56)
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 3
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.